CLINICAL TRIAL: NCT00180154
Title: Tumor Metabolism of Lung Cancer Underwent Percutaneous Radiation Measured With F-18-FDG-PET
Brief Title: Tumor Metabolism of Lung Cancer in Patients Who Underwent Percutaneous Radiation Measured With F-18-FDG-PET
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Jörg Kotzerke, Prof. Dr., Technische Universität Dresden
Other Study IDs: BCA-FDG-FU
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Lung Cancer
Keywords: radiation therapy; F-18-FDG; NSCLC
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to describe the regional and global FDG-kinetics in non-small-cell lung cancer (NSCLC) during percutaneous radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC not curable by surgery
* Karnofsky > 80%
* Tumor volume and localization allow curative radiotherapy
* Written consent

Exclusion Criteria:

* Metastases
* Diabetes
* Pregnancy
* Psychiatric impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes consecutive patients from Department of Radiooncology with inoperable non-small cell lung cancer (NSCLC) intended for a curative radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Kotzerke, MD, Principal Investigator — Department of Nuclear Medicine
Locations (1):
- Department of Nuclear Medicine, Dresden, Germany